CLINICAL TRIAL: NCT03778385
Title: Exercise Specificity and Endogenous Pain Modulation
Brief Title: Influence of Exercise Type, Pain Mechanisms, and Biopsychosocial Contributions to Pain Relief in Those With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marquette University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HR-3035; R15HD090265 (NIH); TL1TR001437 (NIH); UL1TR001436 (NIH)
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Exercise; Pain; Physical Activity; Body Composition
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All subjects will participate in two randomized exercise sessions. Clinical and experimental pain assessment will be performed before, during, and after each exercise task.
Who Masked: Participant
Masking Description: Participants are masked to the primary hypothesis of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric Exercise (Experimental): Submaximal isometric resistance exercise of the arm.
  Interventions: Other: Exercise
- Dynamic Exercise (Experimental): Submaximal dynamic resistance exercise of the arm.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Submaximal exercise is performed in randomized order with the participant seated and the arm supported in an adjustable hand-arm orthosis.

SUMMARY:
The purpose of this study is to investigate the influence different types of exercise, pain mechanisms, and biopsychosocial contributions on how people with and without fibromyalgia report pain. Exercise will be performed with the arm at a submaximal intensity. Participants will undergo a variety of pain assessments, including clinical questionnaires and pain perception. This study will improve our understanding of how people with and without fibromyalgia respond to different resistance exercise types and whether physical activity and body composition has an influence on the response.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic widespread pain condition that is mostly prevalent in middle-aged women. Exercise is one of the few therapies that can alleviate fibromyalgia symptoms. Despite exercise being a major component of rehabilitation, exercise guidelines are unclear, often leading to symptom exacerbation and low compliance. Previous research has demonstrated that women with fibromyalgia may have different post-exercise pain responses when undergoing an exercise task. Factors critical to optimal exercise prescription are not known, including the most effective type of exercise, mechanisms responsible for pain relief, and biopsychosocial influences. This study investigates the use of exercise as a nonpharmacological pain management tool for people with fibromyalgia.

The purpose of this study is to investigate the acute exercise-induced pain response after isometric and dynamic muscle contractions in people with and without fibromyalgia. All participants will attend up to three sessions with approximately one week between sessions at a metropolitan university laboratory setting. Participants will perform different types of submaximal exercise for a maximum of ten minutes and complete pain assessments each session. Pain and psychosocial influences are measured with multiple established clinical questionnaires. Pressure pain sensitivity is tested by application of a mechanical stimulus to the arms and legs. To investigate a participant's innate ability to inhibit pain, the mechanical stimulus will be assessed with and without limb submersion in a cold-water bath. Physical activity is measured via questionnaire and use of activity monitors, while body composition is measured with a dual energy x-ray absorptiometry scan.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia
* Healthy Controls without fibromyalgia
* Stable medical management plan for four weeks prior to participation in the study.
* Physical Activity Readiness Questionnaire (PAR-Q)
* English proficiency

Exclusion Criteria:

* Elbow arthritis
* Carpal tunnel syndrome
* Cervical surgery
* Cerebrovascular accident / stroke
* Multiple sclerosis
* Parkinson's disease
* Any central neurodegenerative disease
* Traumatic brain injury
* Peripheral neuropathy of the upper extremity
* Myocardial infarction
* Chronic obstructive pulmonary disease
* Any unstable medical or psychiatric condition
* Diabetes mellitus
* Active cancer
* Lymphedema of the upper extremity
* Claustrophobia
* Raynaud's phenomenon
* Osteoporosis
* Major depressive disorder
* Bipolar disorder
* Rheumatoid arthritis
* Lupus
* Polymyalgia rheumatica
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Short-Form McGill Pain Questionnaire to 7-days after performance of exercise. | Before and up to 7-days after performance of exercise.
  The Short-Form McGill Pain Questionnaire is a multi-dimensional tool to assess pain quality in chronic pain patients. Participants rate the intensity of pain and related symptoms they felt during the past week on 0 to 3 scale, with 0 being no pain and 3 being severe. The total score ranges from a minimum of 0 to maximum 45 with higher scores indicating worse symptoms.
Change from Baseline Fibromyalgia Impact Questionnaire to 7-days after performance of exercise. | Before and up to 7-days after performance of exercise.
  The Fibromyalgia Impact Questionnaire - Revised measures function, overall impact, and symptoms of fibromyalgia. Participants rate the difficulty in performing daily tasks, the impact of their symptoms, and intensity of fibromyalgia symptoms on a 0 to 10 scale, with 10 signifying greater significance. The total score ranges from a minimum of 0 to maximum of 210 with higher scores indicating worse function and symptoms.
Change from Baseline Pain Rating from a Pressure Pain Device to immediately after performance of exercise. | Before and immediately after performance of exercise.
  Application of mechanical stimulus through a weighted Lucite edge will be applied to the finger for a maximal duration of 2 minutes. Subjects will provide a pain rating every 20 seconds during the 2-minute test. Pain ratings are provided with use of a Numerical Pain Rating Scale that ranges from 0 (no pain) to 10 (worst pain).
Change from Baseline Pressure Pain Threshold to immediately after performance of exercise. | Before and immediately after exercise.
  Application of a pressure stimulus is applied to the bicep muscle and quadriceps muscle at a rate of 50kPa per second until the pressure first becomes painful.
Change from Baseline Numerical Pain Rating Scale to 7-days after performance of exercise. | Before, during, and up to 7-days after performance of exercise.
  Pain in the exercising limb and whole body will be reported. Pain ratings are provided with use of a Numerical Pain Rating Scale that ranges from 0 (no pain) to 10 (worst pain).
Change in Pain Catastrophizing before to after exercise. | Through study completion, an average of 3 weeks.
  Measures the exaggerated negative mental set brought to bear during an actual or anticipated painful experience. Measured with the Pain Catastrophizing Scale which has subscales of rumination, magnification, and helplessness. Rumination scale ranges from 0 to 16 with higher score indicating higher levels of rumination. Magnification scale ranges from 0 to 12 with higher scores indicating higher levels of magnification. Helplessness scale ranges from 0 to 24 with higher scores indicating higher levels of helplessness. The subscale scores are summed to compute a total score ranging from 0 to 52 with higher scores indicating higher levels of pain catastrophizing.
Baseline Tampa Scale of Kinesiophobia - 11 | At the beginning of each session.
  Measures pain-related fear in relation to movement or avoidance type behaviors. A total score is computed ranging from 0 to 44 with higher scores indicating higher levels of pain-related fear.
Change from Baseline PROMIS Short Form v1.0 - Fatigue 7a at completion of study. | At the beginning of each exercise session.
  Measures the experience and impact of fatigue on daily activity. The PROMIS Short Form v1.0 - Fatigue 7a measures subjective feelings of tiredness to a sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Participants rank the level of tiredness on a scale of 1 (never) to 5 (always). The total score ranges from 7 to 35 with 35 indicating greater levels of exhaustion that impacts ability to perform daily tasks.
American College of Rheumatology Diagnostic Criteria for Fibromyalgia | At the beginning of each session.
  Questionnaire characterizing the symptoms of those with fibromyalgia. The scale is composed of 3 subscales; widespread pain index, symptom severity score A and B. The widespread pain index ranges from 0 to 19 with 19 indicating greater number of body areas in which pain was experienced. The symptom severity score A ranges from 0 to 9 with 9 indicating greater symptom severity. The symptom severity score B ranges from 0 to 3 with 3 indicating greater number of symptoms experienced. The total Symptom Severity Score is calculated by adding symptom severity score A and symptom severity score B with a total range of 0 (no symptoms) to 12 (great deal of symptoms).
Conditioned Pain Modulation | Day 1 of enrollment
  The difference in pressure pain (measured via pressure algometry) at the biceps and quadriceps with and without the subject's limb placed in an ice water bath.
Physical Activity Assessment Tool | Up to 7 days.
  The Physical Activity Assessment Tool estimates the amount of physical activity performed and perceptions towards participation in physical activity. The total amount of time per day (minutes/day) is calculated for time spent in moderate to vigorous physical activity. With 0 minutes indicating no time spent in moderate to vigorous physical activity and higher values indicating greater time spent in moderate to vigorous physical activity.
Total time spent in sedentary and moderate to vigorous physical activity measured by an Actigraph wGT3x over the course of 7 days. | Worn continuously for a 7-day period during study enrollment.
  An Actigraph wGT3x is a wrist worn device that is used to track the amount and intensity of physical activity performed over the course of seven days. Total time spent in sedentary and moderate to vigorous physical activity is measured in minutes.
Baseline Lean Mass | 7 to 14 days after enrollment.
  Measurement of lean mass with use of dual energy x-ray absorptiometry testing.
Baseline Fat Mass | 7 to 14 days after enrollment.
  Measurement of fat mass with use of dual energy x-ray absorptiometry testing.

SECONDARY OUTCOMES:
Change from Baseline Maximal Voluntary Force to immediately after performance of exercise. | Before and immediately after performance of exercise.
  Maximal force produced with the arm when performing a bending motion of the elbow. Maximal torque is measured with an isokinetic dynamometer with higher levels indicating greater amount of force.
Baseline voluntary muscle activation of the biceps muscle | Through study completion, an average of 3 weeks.
  Assess each subject's ability to voluntarily activate their bicep muscle when performing a maximal voluntary contraction of the elbow flexors. Participants will generate maximal force from their elbow flexors with application of muscle stimulation. Muscle stimulation is provided via electrodes placed on the skin overlying the biceps muscle and activation of the muscle will be achieved by a constant-current stimulator. Force is recorded via isokinetic dynamometry. To assess voluntary activation, a single twitch will be interpolated during the plateau of the maximal voluntary contraction force by the stimulator.
Change from Baseline Heart Rate to immediately after performance of exercise. | Measured before, during, and immediately after exercise.
  Heart rate is measured with an automated cuff applied to the wrist.
Change from Baseline Blood Pressure to immediately after performance of exercise. | Measured before, during, and immediately after exercise.
  Blood pressure is measured with an automated cuff applied to the wrist.
Change from Baseline Rating of Perceived Exertion to immediately after performance of exercise | Measured before, during, and immediately after exercise.
  Rating of Perceived Exertion refers to the total amount of exertion a participant is feeling and measured with a modified BORG scale ranging from 0 (nothing) to 10 (maximal exertion).
Baseline sensory threshold assessed with von Frey monofilaments | At the beginning of each session.
  Monofilaments will be applied perpendicular to the skin in ascending order, the lowest-size filament to induce sensation is recorded.
Change from baseline pain unpleasantness up to 7 days after exercise. | Before, during, and up to 7-days after performance of exercise.
  Unpleasantness in the exercising limb will be reported with a 0-10 numerical rating scale.
Change from baseline PROMIS Short Form v1.0 Pain Interference 6b up to 7 days after exercise. | Before, during, and up to 7-days after performance of exercise.
  A 6-item questionnaire will help measure interference of pain on functional daily activity.

CONTACTS AND LOCATIONS:
Overall Officials: Marie K Hoeger Bement, PT, PhD, Principal Investigator — Marquette University
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Berardi G, Eble C, Hunter SK, Bement MH. Localized Pain and Fatigue During Recovery From Submaximal Resistance Exercise in People With Fibromyalgia. Phys Ther. 2023 Jun 5;103(6):pzad033. doi: 10.1093/ptj/pzad033. PMID 37384640